CLINICAL TRIAL: NCT01399216
Title: Effects of a Supplement Containing Fucoidan as a Major Component on Basal Body Temperature: a Placebo Controlled, Cross-over Study
Brief Title: Effects of a Supplement Containing Fucoidan on Basal Body Temperature
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hiroshima University (Other)
Collaborators: Three Peace Co., Ltd., Japan (Unknown)
Responsible Party: Principal Investigator, Fumiko Higashikawa, Associate Professor, Hiroshima University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Prevention
Other Study IDs: eki-420
Record Dates: First submitted 2011-07-19; First posted 2011-07-21 (Estimated); Last update posted 2012-12-17 (Estimated); Status verified 2012-12

CONDITIONS: Low Basal Body Temperature

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fucoidan supplement (Experimental)
  Interventions: Dietary Supplement: Supplement containing fucoidan, EPA, and DHA
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Supplement containing fucoidan, EPA, and DHA — 75 mg fucoidan per day, for 8 weeks
  Arms: Fucoidan supplement
Dietary Supplement: Placebo — for 8 weeks
  Arms: Placebo

SUMMARY:
We aim to determine whether a supplement containing fucoidan isolated from Mekabu (sporophyll of Undaria pinnatifida), EPA, and DHA has effects of elevating basal body temperature in subjects with low basal body temperature.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with basal body temperature < 36.0 ºC
* Healthy as based on medical history and physical examination
* Willing not to donate blood during the study
* Informed consent signed

Exclusion Criteria:

* Renal or hepatic dysfunction
* Heart disease
* Participation in any clinical trial within 90 days of the commencement of the trial
* Subjects who are taking medicines or functional food that may affect basal body temperature

Ages: 55 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 19 (Actual)
Dates: Start 2011-07; Primary Completion 2012-03 (Actual); Study Completion 2012-03 (Actual)

PRIMARY OUTCOMES:
Basal body temperature | up to 20 weeks

SECONDARY OUTCOMES:
Change from baseline in serum lipid levels (total cholesterol, LDL cholesterol, HDL cholesterol, and triglyceride) | Weeks 0, 8, 12, and 20

CONTACTS AND LOCATIONS:
Overall Officials: Fumiko Higashikawa, PhD, Principal Investigator — Hiroshima University
Locations (1):
- Hiroshima University, Hiroshima, Japan